CLINICAL TRIAL: NCT02876861
Title: Neoadjuvant Chemotherapy Versus Surgery Alone in Patients With High-Grade Upper Tract Urothelial Carcinoma
Brief Title: Neoadjuvant Chemotherapy Versus Surgery Alone in Patients With High-Grade UTUC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Central South University (Other); The Third Xiangya Hospital of Central South University (Other); Hunan Cancer Hospital (Other); Hunan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYURO001
Record Dates: First submitted 2016-08-14; First posted 2016-08-24 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2022-06

CONDITIONS: High-Grade Upper Tract Urothelial Carcinoma
Keywords: Neoadjuvant chemotherapy; upper tract urothelial carcinoma
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery alone (Active Comparator): Surgeons: the operation shall be performed by senior urologic surgeons. Try to achieve the consistency of operation quality.
  Operation: Radical nephroureterectomy (RNU) with an ipsilateral bladder cuff or distal ureterectomy.
  Interventions: Procedure: Radical nephroureterectomy; Procedure: Distal ureterectomy
- Neoadjuvant chemotherapy and Surgery (Experimental): Experimental: Neoadjuvant chemotherapy group
  Neoadjuvant chemotherapy(Gemcitabine and Cisplatin):
  Gemcitabine, 1250mg/m2, d1 d8, Cisplatin, 75mg/m2, d1-d3, 21d, 2-4 cycles.
  Surgery:
  2-3weeks after Neoadjuvant chemotherapy
  Surgeons: the operation shall be performed by senior urologic surgeons. Try to achieve the consistency of operation quality.
  Operation: Radical nephroureterectomy (RNU) with an ipsilateral bladder cuff or distal ureterectomy.
  Interventions: Procedure: Radical nephroureterectomy; Procedure: Distal ureterectomy; Drug: Neoadjuvant Chemotherapy

INTERVENTIONS:
Procedure: Radical nephroureterectomy — Radical nephroureterectomy (RNU) with an ipsilateral bladder cuff
Procedure: Distal ureterectomy — Distal ureterectomy.
Drug: Neoadjuvant Chemotherapy — Gemcitabine, 1250mg/m2, d1 d8, Cisplatin, 75mg/m2, d1-d3, 21d, 2-4 cycles.
  Other Names: GC
  Arms: Neoadjuvant chemotherapy and Surgery

SUMMARY:
The purpose of this study is to see if getting chemotherapy with Gemcitabine and Cisplatin (GC) for 2-4 cycles can help shrink the tumor before undergoing surgery and improves the overall survival for high-grade upper tract urothelial carcinoma.

DETAILED DESCRIPTION:
The purpose of this study is to see if getting chemotherapy with Gemcitabine and Cisplatin (Gemcitabine, 1250mg/m2, d1 d8, Cisplatin, 75mg/m2, d1-d3, 21d, 2-4 cycles) for 2-4 cycles can help shrink the tumor before undergoing surgery and improves the overall survival for high-grade upper tract urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade upper tract transitional cell carcinoma at MSKCC or a participating site and/or radiographically visible tumor stage T2-T4a N0/X M0 disease with positive selective urinary cytology. Hydronephrosis associated with tumor on imaging or biopsy will be considered invasive by definition.
* Medically appropriate candidate for radical nephroureterectomy or ureterectomy as per MSKCC or a participating site attending urologic oncologist
* Karnofsky Performance Status ≥ 70%
* Age ≥ 18 years of age
* Required Initial Laboratory Values:

Absolute neutrophil count ≥ 1500 cells/mm3 Platelets ≥ 100,000 cells/mm3 Hemoglobin ≥ 9.0g/dL Bilirubin ≤ 1.5 Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN for the institution Alkaline phosphatase ≤ 2.5 x upper limit of normal (ULN) for the institution Serum creatinine ≤ 1.5 mg/dL and calculated creatinine clearance ≥ 55 If female of childbearing potential, serum pregnancy test is negative.

* Patients with reproductive potential must use an effective method to avoid pregnancy for the duration of the trial.

ml/min/1.73m2 using the formula: Chronic kidney disease (CKD) epi : glomerular filtration rate (GFR) = 141 X min(Scr/κ,1)α X max(Scr/κ,1)-1.209 X 0.993 Age X 1.018 [if female] X 1.159 [if black]

* Scr is serum creatinine, k is 0.7 for females and 0.9 for males, a is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/k or 1, and max indicates the maximum of Scr/k or 1.
* If female of childbearing potential, serum pregnancy test is negative.
* Patients with reproductive potential must use an effective method to avoid pregnancy for the duration of the trial

Exclusion Criteria:

* Concomitant bladder urothelial carcinoma is acceptable if it is organ confined and surgically resectable.
* Presence of carcinoma in situ (CIS)
* Prior systemic chemotherapy (prior intravesical therapy is allowed)
* Prior radiation therapy to the bladder
* Evidence of New York Heart Association (NYHA) functional class III or IV heart disease.
* Serious intercurrent medical or psychiatric illness, including serious active infection.
* Preexisting sensory grade 3 neuropathy
* Major surgery or radiation therapy < 4 weeks of starting study treatment.
* Concomitant use of any other investigational drugs
* Any of the following within the 6 months prior to study drug administration:

myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.

* Ongoing cardiac dysrhythmias of NCI CTCAE Version 4.0 grade ≥ 2.
* Uncontrolled hypertension (>150/100 mmHg despite optimal medical therapy).
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection. Patients with HIV but no evidence of AIDS will be considered candidates.
* Concurrent treatment on another clinical trial involving an intervention which may affect the primary endpoint. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
* Ongoing treatment with therapeutic doses of warfarin or low molecular weight heparin (low dose warfarin up to 2 mg po daily or use of subcutaneous low molecular weight heparin for thromboembolic prophylaxis is allowed).
* Pregnancy or breast-feeding. Patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the MSKCC and participating site PI. Male patients must be surgically sterile or agree to use effective contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-02; Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  Disease-free survival

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | after neoadjuvant chemotherapy completion, assessed up to 4 weeks
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1
Overall survival (OS) | From date of surgery until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 100 months death from any cause, whichever came first, assessed up to 100 months
  Overall survival
Number of participants with chemotherapy-related adverse events as assessed by National Cancer Institute Common Toxicity Criteria version 4.0. | Through neoadjuvant chemotherapy completion, assessed up to 4 weeks
  Number of participants with chemotherapy-related adverse events as assessed by National Cancer Institute Common Toxicity Criteria version 4.0.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Long Wang, M.D. Ph.D., Study Chair — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South Univeristy, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided